CLINICAL TRIAL: NCT05814172
Title: Beijing Tongren Hospital, Capital Medical University
Brief Title: ADL and CONUT for Predicting 1-year Mortality Risk in Older Adults After Hip Fracture
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TREC2023-KY026
Record Dates: First submitted 2023-03-19; First posted 2023-04-14 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-03

CONDITIONS: All-cause Mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Death by 1 y: patients who dieded within 1-year after discharge due to hip fracture surgery
  Interventions: Other: no intervention
- Alive at 1 y: patients who survived 1-year after discharge due to hip fracture surgery
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Hip fracture has a serious impact on the quality of life and even the survival of older adults. The multidisciplinary management of hip fracture has been shown to be effective in improving patient outcome and cost-effective in international studies. As geriatricians and members of a multi-disciplinary team（MDT）, we are aware of various scores in predicting the 1-year mortality risk in hospitalized older adults with multimorbidity. However, given the need for a deeper understanding of the preoperative status of elderly patients who were suffering from pain, tension, anxiety, delirium,etc., we hope to explore a simple, quick, objective, and accurate method for assessing the status of elderly patients with hip fractures to predict their survival risk.

DETAILED DESCRIPTION:
This was a single-center retrospective cohort study which were approved by the Clinical Research Ethics Committee of Beijing Tongren Hospital, Capital Medical University (TREC2023-KY026). Demographic characteristics and medical parameters, such as age, gender, body mass index (BMI), comorbidities, hemoglobin , lymphocytes, C-reactive protein (CRP), fasting blood glucose, creatinine, total protein, albumin, triglycerides, total cholesterol and American Association of Anesthesiologists (ASA) were collected from the electronic medical record system. Controlling nutritional status (CONUT) was calculated from 3 variables: serum albumin concentration, total cholesterol concentration, and lymphocyte count, as previously reported. All enrolled patients were followed-up in an outpatients setting. Survival data were obtained via direct contact with patients or patients' caregiver by their physicians at the hospital , or via telephone interview of their family by dedicated coordinators and investigators. The follow-up lasted for one year and the last follow-up was ended on December 31, 2022. All analyses were performed using SPSS version 19.0 (SPSS, Chicago, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

1. patients aged ≧65 years old;
2. patients diagnosed with hip fracture, including femoral neck fracture, femoral intertrochanteric fracture, and femoral subtrochanteric fracture;
3. patients whose injury was within 21 days of presentation.

Exclusion Criteria:

1. patients aged <65 years old;
2. patients with pathological fractures due to tumor metastasis or infection or inherited bone disorder;
3. patients with avascular necrosis of femoral head;
4. patients with periprosthetic fractures;
5. old fracture patients treated more than 21 days from injury;
6. patients with severe trauma or fracture in other parts;
7. patients and their families who could not bear the surgical risk and are unwilling to receive surgical treatment;
8. patients died in hospital.

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older adults with unilateral hip fractures who received surgical treatment in our hospital from January 2014 to December 2021 were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 303 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Mortality | Calculated from the time of discharge, each patient was followed up 1 year, all-cause death in 1 year after discharge was counted.
  After discharge, all enrolled patients were followed-up in an outpatients setting. Survival data were obtained via direct contact with patients or patients' caregiver by their physicians at the hospital , or via telephone interview of their family by dedicated coordinators and investigators. Survival data were obtained via direct contact with patients or patients' caregiver by their physicians at the hospital , or via telephone interview of their family by dedicated coordinators and investigators. Outcomes were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: QI LIU, Study Director — Beijing Tongren Hospital
Locations (1):
- Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided